CLINICAL TRIAL: NCT05209035
Title: Randomized-Controlled Trial of Trazodone on Reducing Plasma sST2 Level and Neurodegeneration Progression in Patients With Amnestic Mild Cognitive Impairment and Obstructive Sleep Apnea
Brief Title: Evaluation of Trazodone in OSA-MCI
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hong Kong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Timothy Kwok, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021.038
Record Dates: First submitted 2022-01-13; First posted 2022-01-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment; Obstructive Sleep Apnea
MeSH Terms: conditions — Cognitive Dysfunction; Sleep Apnea, Obstructive | interventions — Trazodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trazodone (Active Comparator)
  Interventions: Drug: Trazodone
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Trazodone — Trazodone 50mg daily
  Arms: Trazodone
Other: Placebo — Starch 50mg
  Arms: Placebo

SUMMARY:
Alzheimer's disease (AD) is a progressive and multifactorial neurodegenerative disease. Before progressing to AD, individuals may experience mild cognitive impairment (MCI). While these individuals with MCI have an increased risk of progressing to AD, emerging studies reveal that obstructive sleep apnea (OSA) is a risk factor for both MCI an well as AD. Thus, it is worthwhile to identify clinical management or interventions that retard the conversion of subjects with comorbid MCI and OSA and AD.

A randomized, double-blind, placebo-controlled study proposed herein aims to examine the effect of trazodone on reducing level sST2 and protein markers that are associated with neurodegeneration in the plasma of subjects with comorbid OSA and MCI. In this 1-year study, 124 study participants will undergo a series of neurocognitive assessments.

ELIGIBILITY:
Inclusion Criteria:

* Able to swallow trazodone capsules
* Stable pharmacological treatment of any other chronic conditions for at least 30 days prior to screening
* A diagnosis of mild cognitive impairment (MCI)
* A diagnosis of obstructive sleep apnea (OSA), and Apnea-Hypopnea Index > 5
* Neuroimaging obtained during screening consistent with a clinical diagnosis of Alzheimer's disease (AD) and without findings of significant exclusionary abnormalities
* Written informed consent to participate in the study provided by the patient

Exclusion Criteria:

* Diagnosis of dementia, neurodegenerative condition, seizure disorder or other infectious, metabolic, or systemic disease affecting the central nervous system
* Vitamin B12 or folate deficiency
* Diagnosis of mental health disorders
* Nootropic drugs except for AD prescriptions stable for at least 30 days
* Suspected or known allergy to trazodone
* Intake of drugs or substances potentially involved in clinically significant inhibition or induction of CYP34A or P-gp-medicate drug interactions with trazodone within 4 weeks or 5 half-lives of the interacting drug prior to administration of trazodone and throughout the course of the study
* Previous exposure to anti-Aβ vaccines
* Concurrent treatment with antipsychotic agents, antiepileptics centrally active antihypertensive drugs, sedatives, opioids, mood stabilizers, or benzodiazepines within 4 weeks of screening visit
* Patients who are receiving non-benzodiazepine hypnotics
* Clinically significant, advanced, or unstable disease that might interfere with outcome evaluations

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-05-10 (Actual); Primary Completion 2025-05-02 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
sST2 | Baseline, Week 4, 13, 26 and 52
  The change of plasma sST2 levels
Clinical Dementia Rating Score | Baseline, Week 26 and 52
  The change in Clinical Dementia Rating global score

CONTACTS AND LOCATIONS:
Overall Officials: Timothy CY Kwok, Principal Investigator — Chinese University of Hong Kong; Susanna Ng, Principal Investigator — Chinese University of Hong Kong; Nancy Ip, Principal Investigator — The Hong Kong University of Science and Technology
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong